CLINICAL TRIAL: NCT00377832
Title: Acetaminophen for Fetal Tachycardia: a Randomized Pilot Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment and lack of funding
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0605008549; 4730406 (Other: New York Hospital Queens IRB)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Fever; Heart Rate, Fetal (FHR)
Keywords: Fetal tachycardia; Fever in labor; Acetaminophen; Non reassuring fetal status
MeSH Terms: conditions — Fever | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Active Comparator): Acetaminophen 975 mg once
  Interventions: Drug: Acetaminophen 975 mg

INTERVENTIONS:
Drug: Acetaminophen 975 mg — Acetaminophen 975 mg by mouth once only
  Other Names: Tylenol
  Arms: 2

SUMMARY:
The most common cause of fetal tachycardia is maternal fever. Fetal tachycardia often precedes the maternal fever, and fetal tachycardia confounds the interpretation of electronic fetal monitoring (EFM), increasing the rate of cesarean delivery for non-reassuring fetal status (NRFS). Our hypothesis is that treatment of fetal tachycardia with acetaminophen will significantly lower maternal body temperature and significantly lower baseline fetal heart rate (FHR). The importance is that interpretation of EFM will improve, thus allowing for a decrease in cesarean delivery for NRFS.

DETAILED DESCRIPTION:
This trial is a randomized, non-placebo controlled, assessment of whether acetaminophen can lower maternal temperature and baseline fetal heart rate in laboring patients with fetal tachycardia.

Term singleton cephalic pregnancies in active phase labor (spontaneous or induced) with fetal tachycardia will be recruited. Patient will be excluded for:

* Exclusion criteria (prior to randomization):
* Acetaminophen allergy
* Clinical chorioamnionitis
* Maternal fever
* Non-reassuring fetal status (NRFS), which is the designation for fetal heart rate abnormalities requiring cesarean delivery
* Previous cesarean delivery
* Multifetal gestation
* Breech presentation
* Known fetal anomaly
* Known contraindication to vaginal delivery

Primary outcome measures are:

1. Maternal body temperature (oral) 90 minutes after treatment
2. Baseline FHR

Secondary outcome measures are:

1. Temperature difference before and after treatment
2. Rate of cesarean delivery
3. Rate of determination of NRFS
4. Rate of subsequent development of maternal fever
5. Rate of diagnosis of clinical chorioamnionitis
6. Rate of neonatal sepsis

Power calculation Internal data collection at our institution of 53 patients showed a mean decrease in temperature of patients in labor with fever receiving acetaminophen is 0.3 degrees C measured an average (mean) of 90 minutes after administration of acetaminophen. Mean oral temperature before acetaminophen was 38.32, SD 0.33. Mean oral temperature after acetaminophen was 38.03, SD 0.85.

Sample size calculation shows that 27 patients are needed in each group to show significant difference using alpha 5% and beta 50%.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy
* Singleton pregnancy
* Pregnancy with cephalic presentation
* Pregnancy in active phase labor
* Fetal tachycardia

Exclusion Criteria:

* Acetaminophen allergy
* Clinical chorioamnionitis
* Maternal fever
* Non-reassuring fetal status or fetal heart rate abnormalities requiring cesarean delivery
* Previous cesarean delivery
* Multifetal gestation
* Breech presentation
* Known fetal anomaly
* Known contraindication to vaginal delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Skupski, MD, Principal Investigator — Weill Medical College of Cornell University, New York Hospital Medical Center of Queens
Locations (1):
- New York Hospital Medical Center of Queens, Flushing, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment 9/2006 until 12/2010 13 patients recruited No funding
Pre-assignment Details: All participants included in assigned groups
Period: Overall Study
Arm/Group | In Labor With a Fever Will Give no Medication | In Labor With a Fever Will Get Acetaminophen 975 mg Orallyonce
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Medication | Acetaminophen 975 mg Once | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.4 (3.4) | 26.1 (4.6) | 26.3 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maternal Body Temperature 90 Minutes After Randomization
Description: Fever in labor is identified,consenting and randomization occurs, either acetaminophen is given or no medication is given, then 90 minutes later maternal temperature is recorded.
Time Frame: 90 minutes
Measure: Median (Inter-Quartile Range); unit: degrees centigrade
Arm/Group | In Labor With a Fever Will Give no Medication | In Labor With a Fever Will Get Acetaminophen 975 mg Orallyonce
Number analyzed (Participants) | 7 | 6
degrees centigrade | 38 [37.3 to 38.5] | 37.4 [37.1 to 37.8]

2. Primary Outcome: Baseline Fetal Heart Rate (FHR) After Treatment
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | No Medication | Acetaminophen 975 mg Once
Number analyzed (Participants) | 7 | 6
beats per minute | 167.6 (17.5) | 152.5 (9.4)

3. Secondary Outcome: Temperature Difference Before and After Treatment
Description: Maternal temperature difference before randomization and 90 minutes after randomization in degrees Centigrade
Time Frame: 90 minutes
Measure: Median (Inter-Quartile Range); unit: degrees Centigrade
Arm/Group | In Labor With a Fever Will Give no Medication | In Labor With a Fever Will Get Acetaminophen 975 mg Orallyonce
Number analyzed (Participants) | 7 | 6
degrees Centigrade | 0.3 [-0.6 to 1.6] | -0.15 [-0.4 to 0.1]

4. Secondary Outcome: Rate of Cesarean Delivery
Description: Rate of cesarean delivery
Time Frame: Labor--up to 24 hours
Measure: Number; unit: participants
Arm/Group | In Labor With a Fever Will Give no Medication | In Labor With a Fever Will Get Acetaminophen 975 mg Orallyonce
Number analyzed (Participants) | 7 | 6
participants | 1 | 2

5. Secondary Outcome: Rate of Determination of Non-reassuring Fetal Status
Description: Non-reassuring fetal status is when cesarean delivery or operative vaginal delivery (forceps or vacuum) are performed for fetal heart rate abnormalities.
Time Frame: Labor--up to 24 hours
Measure: Number; unit: participants
Arm/Group | In Labor With a Fever Will Give no Medication | In Labor With a Fever Will Get Acetaminophen 975 mg Orallyonce
Number analyzed (Participants) | 7 | 6
participants | 1 | 2

6. Secondary Outcome: Rate of Subsequent Development of Maternal Fever
Description: Rate of subsequent development of maternal fever, i.e., the number of participants who developed fever.
Time Frame: Labor--up to 24 hours
Measure: Number; unit: participants
Arm/Group | In Labor With a Fever Will Give no Medication | In Labor With a Fever Will Get Acetaminophen 975 mg Orallyonce
Number analyzed (Participants) | 7 | 6
participants | 6 | 2

7. Secondary Outcome: Rate of Diagnosis of Clinical Chorioamnionitis
Description: Rate of diagnosis of clinical chorioamnionitis, i.e., the number of participants who developed chorioamnionitis.
Time Frame: Labor--up to 24 hours
Measure: Number; unit: participants
Arm/Group | In Labor With a Fever Will Get no Medication | In Labor With a Fever Will Get Acetaminophen 975 mg Orallyonce
Number analyzed (Participants) | 7 | 6
participants | 1 | 0

8. Secondary Outcome: Rate of Neonatal Sepsis
Description: the number of participants who developed neonatal sepsis
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | In Labor With a Fever Will Give no Medication | In Labor With a Fever Will Get Acetaminophen 975 mg Orallyonce
Number analyzed (Participants) | 7 | 6
participants | 0 | 0

ADVERSE EVENTS:
Groups:
- No Medication: In labor, fever is identified, consent and randomization occurs, then no medication is given.
- Acetaminophen 975 mg Once: In labor, fever is identified, consent and randomization occurs, then acetaminophen is given.
Arm/Group | No Medication | Acetaminophen 975 mg Once
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Poor recruitment and lack of funding led to early termination of the trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No